CLINICAL TRIAL: NCT02914938
Title: A Three-Arm Study of ME-401 Monotherapy in Subjects With Relapsed/Refractory CLL, SLL, or FL, of ME-401 in Combination With Rituximab in Subjects With Relapsed/Refractory CLL/SLL or B-cell NHL, and of ME-401 in Combination With Zanubrutinib in Subjects With Relapsed/Refractory CLL/SLL or B-cell NHL
Brief Title: A Study of ME-401 in Subjects With CLL/SLL, FL, and B-cell Non Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: discontinuation of zandelisib program
Sponsor: MEI Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ME-401-002
Record Dates: First submitted 2016-09-12; First posted 2016-09-26 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2022-12

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL); Follicular Lymphoma (FL); Marginal Zone B Cell Lymphoma; Diffuse Large B-cell Lymphoma (DLBCL); High Grade Non-Hodgkin's Lymphoma; Mantle Cell Lymphoma (MCL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell | interventions — ME-401; Rituximab; zanubrutinib

STUDY DESIGN:
Intervention Model Description: This is a three-arm study of ME-401 alone, of ME-401 in combination with rituximab, and of ME-401 in combination with zanubrutinib in subjects with relapsed/refractory CLL/SLL or B cell NHL. The 3 arms of the study will be conducted in parallel, with subject allocation to ME 401 alone, ME-401 plus rituximab, or ME 401 plus zanubrutinib based on disease type and availability of an open enrollment slot.
Oversight: Data Monitoring Committee: No

ARMS (3):
- ME-401 Alone (Experimental): This arm is an open-label, dose escalation study to determine the safety, efficacy and pharmacokinetics of ME-401 along with the mBED, MTD, and DLTs. There are 4 planned cohorts which may enroll up to 61 subjects.
  Interventions: Drug: ME-401
- ME-401 in Combination with Rituximab (Experimental): The second arm is an open label study to evaluate the safety, efficacy, and pharmacokinetics of ME-401 in combination with rituximab in subjects with various B-cell malignancies. There are two planned cohorts which may enroll up to 30 subjects.
  Interventions: Drug: ME-401; Drug: Rituximab
- ME-401 in Combination with Zanubrutinib (Experimental): The third arm is an open label study evaluating the safety, efficacy, MTD, DLT and pharmacokinetics of ME-401 in combination with zanubrutinib in subjects with various B-cell malignancies. This arm will include 2 stages: a safety evaluation stage (cohort of 6-12 subjects) and a disease-specific expansion cohort stage (up to 74 subjects).
  Interventions: Drug: ME-401; Drug: Zanubrutinib

INTERVENTIONS:
Drug: ME-401 — 60 mg
Drug: Rituximab — IV infusion 375 mg/m2
  Other Names: Rituxan
  Arms: ME-401 in Combination with Rituximab
Drug: Zanubrutinib — 80 and 160 mg bid
  Arms: ME-401 in Combination with Zanubrutinib

SUMMARY:
A Three-Arm Study of ME-401 in Subjects with Relapsed/Refractory CLL/SLL or FL, of ME-401 in Combination with Rituximab in Subjects with Relapsed/Refractory CLL/SLL or B-cell NHL, and of ME-401 in Combination with Zanubrutinib in Subjects with Relapsed/Refractory CLL/SLL or B-cell NHL

DETAILED DESCRIPTION:
This is a three-arm study of ME-401 alone, of ME-401 in combination with rituximab, and of ME-401 in combination with zanubrutinib in subjects with relapsed/refractory CLL/SLL or B cell NHL. The 3 arms of the study will be conducted in parallel, with subject allocation to ME-401 alone, ME-401 plus rituximab, or ME-401 plus zanubrutinib based on disease type and availability of an open enrollment slot.

ELIGIBILITY:
Inclusion Criteria MEI-401 Alone:

* Diagnosis of relapsed/refractory CLL and/or relapsed/refractory SLL or FL
* No prior therapy with PI3Kd inhibitors
* No prior therapy with Bruton tyrosine kinase (BTK) inhibitors unless the subject was intolerant of BTK therapy or subject had disease progression
* Subjects with CLL/SLL must have prior treatment with BTK inhibitor and must have had progression or recurrence while on treatment of within 12 mos from BTK treatment
* Subject must have failed at least 1 prior systemic therapy
* QT-interval corrected according to Fridericia's formula (QTcF) ≤ 450 milliseconds (ms)
* Left ventricular ejection fraction > 50%
* For subjects, except those with CLL, must have at least one bi-dimensionally measurable nodal lesion >1.5 cm, as defined by Lugano Classification
* Willingness to participate in collection of pharmacokinetic samples
* A negative serum pregnancy test within 14 days of study Day 0, for females of childbearing potential

Inclusion Criteria ME-401 in Combination with Rituximab

* Diagnosis of relapsed/refractory CLL SLL or FL, MZL, DLBCL and high-grade B-cell lymphoma. Subjects must meet the following criteria for relapsed or refractory disease:
* No prior therapy with PI3Kδ inhibitors
* No prior therapy with Bruton tyrosine kinase (BTK) inhibitors unless the subject was intolerant of BTK therapy or subject had disease progression
* Subjects with CLL, SLL, FL, and MZL must have a failure of at least 1 prior systemic therapy and be considered by the investigator a candidate for therapy with a rituximab-based regimen; subjects with DLBCL and high-grade B-cell lymphoma must have a failure of at least 2 prior therapies.
* QT-interval corrected according to Fridericia's formula (QTcF) ≤450 milliseconds (ms)
* Left ventricular ejection fraction > 50%
* For subjects, except those with CLL, must have at least one bi-dimensionally measurable nodal lesion >1.5 cm, as defined by Lugano Classification
* Willingness to participate in collection of pharmacokinetic samples
* A negative serum pregnancy test within 14 days of study Day 0 for females of childbearing potential

Inclusion Criteria ME-401 in Combination with Zanubrutinib

* Diagnosis of relapsed/refractory CLL or histologically-confirmed relapsed/refractory SLL or FL, MZL, MCL, DLBCL NOS (germinal center B-cell type or activated B-cell type)
* No prior therapy with PI3Kδ inhibitors
* No prior therapy with BTK inhibitors
* Subjects with CLL, SLL, FL, MCL, and MZL must have a failure of at least 1 prior systemic therapy, require treatment in the opinion of the investigator, and be considered by the investigator a candidate for therapy subjects with DLBCL and high-grade B-cell lymphoma must have a failure of at least 2 prior therapies
* For subjects with SLL, FL, MZL, MCL, DLBCL: At least one bi dimensionally measurable nodal lesion > 1.5 cm in its longest diameter by CT scan or MRI
* QT-interval corrected according to Fridericia's formula (QTcF) ≤ 450 milliseconds (msec)
* Left ventricular ejection fraction > 50% as measured by echocardiogram or multigated acquisition (MUGA) scan
* Willingness to participate in collection of pharmacokinetic samples
* For females of childbearing potential, a negative serum pregnancy test within 14 days of study Day 0

Exclusion Criteria:

* Known histological transformation from CLL to an aggressive lymphoma
* Uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia
* Subjects who have tested positive for hepatitis B surface antigen and/or hepatitis B core antibody
* Positive for hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody
* Ongoing drug-induced pneumonitis
* History of clinically significant cardiovascular abnormalities
* History of severe bleeding disorders (ME-401 plus zanubrutinib arm only)
* Known central nervous system (CNS) hemorrhage or stroke within 6 months prior to start of study drugs (ME-401 plus zanubrutinib arm only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2016-10; Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Minimum Biologically Effective Dose (mBED) of ME-401 alone | 1 year
  The mBED will be defined as the dose that is safe and that achieves an objective response rate that is not less than 30%.
Maximally Tolerated Dose (MTD) of ME-401 alone | 1 year
  The MTD will be determined as the maximum dose that is safe. DLT rate closest to .25 and not to exceed 2 DLTs in 6 subjects
Dose Limiting Toxicities (DLTs) of ME-401 alone | within the first 56 days
  DLTs will be measured by the number of treatment related AEs that occur within the first 56 days of ME-401 administration, is considered clinically significant by the P.I. and occurs in the presence of supportive care
Evaluate the safety and tolerability of ME-401 plus rituximab | 1 year
  Safety and tolerability will be measured by the number of treatment related AEs
Determine the MTD of ME-401 plus zanubrutinib | 1 year
  The MTD of ME-401 is defined as the dose level with a DLT rate closest to 0.25.
Determine the DLTs of ME-401 plus zanubrutinib | within the first 56 days
  DLTs will be measured by the number of treatment related AEs that occur within the first 56 days of ME-401 plus zanubrutinib
Evaluate the safety and tolerability of ME-401 plus zanubrutinib | 1 year
  Safety and tolerability will be measured by the number of treatment related AEs

SECONDARY OUTCOMES:
Safety profile of ME-401 alone | 1 year
  Safety profile will be measured by number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Efficacy of ME-401 alone as assessed by (OR) | 2 years
  The efficacy of ME-401 alone will be assessed by the overall response (OR) of subjects which is calculated as the percent of subjects achieving complete response (CR), minimal disease negativity (MRD), duration of response (DOR) and progression free survival (PFS).
Evaluate the (AUC) PK of ME-401 alone | 2 years
  Determined by the Area Under the Concentration time curve (AUC)
Evaluate the PK (Cmax) of ME-401 alone | 2 years
  Determined by Peak Plasma Concentration (Cmax)
Efficacy of ME-401 with rituximab | 2 years
  The efficacy of ME-401 with Rituximab will be determined by the overall response (OR) of subjects calculated as the percent of subjects achieving a complete remission (CR), duration of response (DOR) or Progression Free survival (PFS) according to the International Workshop on Chronic Lymphocytic Leukemia (iwCLL)
Evaluate the PK (AUC) of ME-401 with rituximab | 2 years
  Determined by the Area Under the Concentration time curve (AUC)
Evaluate the PK (Cmax) of ME-401 with rituximab | 2 years
  Determined by Peak Plasma Concentration (Cmax)
Efficacy of ME-401 with zanubrutinib | 2 years
  The efficacy of ME-401 with zanubrutinib will be assessed by the overall response (OR) of subjects calculated as the percent of subjects achieving a complete remission (CR), Duration of response (DOR) and progression free survival (PFS)
Evaluate the PK (AUC) of ME-401 in combination with zanubrutinib | 2 years
  Determined by the Area Under the Concentration time curve (AUC)
Evaluate the PK (Cmax) of ME-401 in combination with zanubrutinib | 2 years
  Determined by Peak Plasma Concentration (Cmax)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (23):
  - University of Arizona, Tucson, Arizona
  - Compassionate Care, Corona, California
  - Sylvester Comprehensive Cancer Center (Univ of Miami School of Med), Miami, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber, Boston, Massachusetts
  - Memorial Sloan Kettering, Basking Ridge, New Jersey
  - Memorial Sloan Kettering, Middletown, New Jersey
  - Memorial Sloan Kettering, Montvale, New Jersey
  - Memorial Sloan Kettering, Commack, New York
  - Memorial Sloan Kettering, Harrison, New York
  - NYU Langone Laura & Isaac - Perlmutter Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook, Stony Brook, New York
  - Memorial Sloan Kettering, Uniondale, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Vanderbilt, Nashville, Tennessee
  - University of Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Edmonds, Washington
  - Swedish Cancer Institute, Issaquah, Washington
  - Swedish Cancer Center, Seattle, Washington
  - Carbone Cancer Center, Madison, Wisconsin
- lstituto Oncologico della Svizzera ltaliana Ospedale Regionale Bellinzona e Valli CH, Bellinzona, Switzerland

REFERENCES:
- [Derived] Pagel JM, Soumerai JD, Reddy N, Jagadeesh D, Stathis A, Asch A, Salman H, Kenkre VP, Iasonos A, Llorin-Sangalang J, Li J, Zelenetz AD. Zandelisib with continuous or intermittent dosing as monotherapy or in combination with rituximab in patients with relapsed or refractory B-cell malignancy: a multicentre, first-in-patient, dose-escalation and dose-expansion, phase 1b trial. Lancet Oncol. 2022 Aug;23(8):1021-1030. doi: 10.1016/S1470-2045(22)00333-3. Epub 2022 Jul 11. PMID 35835137